CLINICAL TRIAL: NCT06954233
Title: Voiding, Erectile and Ejaculatory Function After Retroperitoneal Lymph Node Dissection for Testicular Cancer
Brief Title: Voiding and Erectile Function After Retroperitoneal Lymph Node Dissection for Testicular Cancer
Acronym: VEEF-RPLND-TC
Status: Recruiting | Type: Observational
Sponsor: Jagiellonian University (Other)
Responsible Party: Principal Investigator, Anna K. Czech, MD, Principal Investigator, Jagiellonian University
Other Study IDs: VEEF-RPLND-TC
Record Dates: First submitted 2025-04-24; First posted 2025-05-01 (Actual); Last update posted 2025-07-16 (Actual); Status verified 2025-07

CONDITIONS: Testicular Cancer
Keywords: Testicular Cancer; Retroperitoneal Lymph Node Dissection
MeSH Terms: conditions — Testicular Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Adult men with testicular cancer undergoing retroperitoneal lymph node dissection: Adult men with testicular cancer undergoing retroperitoneal lymph node dissection will have uroflowmetry performed and will complete questionnaires focusing on urinary, erectile and ejaculatory function before surgery, after surgery and during 6 months follow-up
  Interventions: Diagnostic Test: Uroflowmetry and questionnaires

INTERVENTIONS:
Diagnostic Test: Uroflowmetry and questionnaires — Uroflowmetry - urine flow assessment Questionnaires: IPSS, ICIQ-MLUTS, IIEF-5, MSHQ-EjD, EQ-5D-5L

SUMMARY:
This study aims to evaluate how retroperitoneal lymph node dissection (RPLND), a surgical treatment for testicular cancer, may affect urinary and sexual functions in men. RPLND involves the removal of lymph nodes from the abdominal area and is sometimes necessary in patients who are not eligible for chemotherapy or who have residual disease after chemotherapy. While this surgery is known to carry a risk of affecting ejaculation, its potential impact on other areas such as urination or erection is not well understood.

The study will prospectively follow adult men undergoing RPLND. It will assess changes in lower urinary tract symptoms, urine flow, ejaculation, erection, and overall quality of life before surgery and during follow-up visits up to 6 months after the operation. Patients will complete standardized questionnaires and undergo simple, non-invasive tests such as urine flow measurement.

By identifying how RPLND may influence urinary and sexual health, this study seeks to improve understanding of the full range of effects of this treatment. The findings may help clinicians better inform patients before surgery and support improved post-operative care.

DETAILED DESCRIPTION:
This is a prospective observational study designed to evaluate the impact of retroperitoneal lymph node dissection (RPLND) on lower urinary tract and sexual function in patients treated for testicular cancer. The study incorporates validated patient-reported outcome measures (PROMs) alongside objective functional assessments to characterize post-RPLND urinary and sexual sequelae over time.

Patients will complete standardized questionnaires preoperatively and at scheduled postoperative intervals, including the International Prostate Symptom Score (IPSS), International Consultation on Incontinence Questionnaire - Male Lower Urinary Tract Symptoms (ICIQ-MLUTS), International Index of Erectile Function (IIEF-5), Male Sexual Health Questionnaire - Ejaculatory Dysfunction (MSHQ-EjD), and EQ-5D-5L for health-related quality of life. Objective evaluation will include uroflowmetry and ultrasound-based measurement of post-void residual volume.

ELIGIBILITY:
Inclusion Criteria:

* Adult male with testicular cancer undergoing retroperitoneal lymph node dissection (RPLND)

Exclusion Criteria:

* History of RPLND
* Lack of consent

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult males with testicular cancer undergoing retroperitoneal lymph node dissection (RPLND)
Sampling Method: Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2025-05-14 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Change in maximal urine flow (Qmax) in uroflowmetry before and after RPLND surgery | 6 months
  Change in maximal urine flow (Qmax) in uroflowmetry before and after RPLND surgery
Change in post-void residual volume (PVR) before and after RPLND surgery | 6 months
  Change in post-void residual volume (PVR) before and after RPLND surgery
Change in total IPSS score before and after RPLND surgery | 6 months
  Patients will complete International Prostate Symptom Score (IPSS) questionnaire to assess urinary function before and after surgery
Change in ICIQ-MLUTS score before and after RPLND surgery | 6 months
  Patients will complete Incontinence Questionnaire - Male Lower Urinary Tract Symptoms - ICIQ-MLUTS questionnaire to assess urinary function before and after surgery

SECONDARY OUTCOMES:
Change in IIEF-5 questionnaire before and after RPLND surgery | 6 months
  Patients will complete International Index of Erectile Function - IIEF-5 questionnaire before and after surgery to assess erectile function
Change in MSHQ-EjD questionnaire before and after RPLND surgery | 6 months
  Patients will complete Male Sexual Health Questionnaire Ejaculatory Dysfunction - MSHQ-EjD questionnaire before and after surgery to assess erectile function

CONTACTS AND LOCATIONS:
Overall Officials: Anna K. Czech, M.D., Principal Investigator — Jagiellonian University
Locations (1):
- Jagiellonian University Medical College, Krakow, Malopolska, Poland

IPD SHARING:
Plan to Share IPD: Undecided